CLINICAL TRIAL: NCT04698928
Title: The Effect of Repetitive Transcranial Magnetic Stimulation on the Cognition in People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chien Tai Hong, Attending physician, Associate Professor, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202004024
Record Dates: First submitted 2020-11-22; First posted 2021-01-07 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease With Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theta burst stimulation group (Experimental): Theta burst stimulation over SMA. 3 section per day, for 5 days, total 15 sections.
  Interventions: Device: Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — Theta burst stimulation over SMA. 3 section per day, for 5 days, total 15 sections.

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease. The cardinal symptoms of PD are tremor, rigidity, bradykinesia and postural instability. Cognitive impairment and dementia are also one of the key features of the non-motor symptoms of PD. At present, the mainstream treatment of PD-dementia is the dopaminergic rivastigmine. Repetitive transcortical magnetic stimulation (rTMS) is a novel non-invasive intervention. Through the magnetic stimulation, brain neurons could be activated by the electrical current. The application of rTMS had been approved by US FDA for the treatment of depression. The possible effect of rTMS may result from the stimulation-related neuronal plasticity. Regarding PD, rTMS also had been found to had some effect on different motor symptoms and cognition. The present study would like to test the accumulative effect of rTMS on cognition of PD. All the study subjects will receive rTMS under intermittent theta burst stimulation (iTBS) mode at supplementary motor area (SMA). Cognitive bahevorial tests and other motor/depression assessments will be assessed before and after the intervention.

DETAILED DESCRIPTION:
The present trial is designed as an open-label, uncontrolled pilot study for evaluating the effect of rTMS on cognitive function in people with Parkinson disease (PD). The primary endpoint is the change of cognitive function, and the secondary endpoint is the improvement of motor symptoms. All participants need to complete the informed consent before they are enrolled into the trial. Preliminary data including age, sex, education, employment, medical history, drug history, disease duration, modified Hoehn-Yahr stage, and UPDRS score are collected. Cognitive function including mini-mental state examination (MMSE), clocking drawing test, Wechsler memory scale (WMS)-world list test and spatial span test, trial making test A and B, category fluency test (animal naming), and beck depression inventory-II are tested by trained neuropsychiatrists. Gait function are evaluated with time up and go (TUG), freezing of gait questionnaire (FOG-Q), and Gait-up device analysis before trial starting. Pre-treatment brain image examined by magnetic resonance image (MRI) and blood sampling for synapse protein level are performed. The participants are then arranged to receive theta burst stimulation for 5 days by using Magstim machine (Super Rapid 2) equipped with air cooled coil (D70), stimulating on supplementary motor area (SMA). After the intervention, post-treatment evaluation including cognition, motor symptoms, gait function, brain MRI, and blood sampling will be performed again with the same methods at 1 month later. Any adverse event during the trial period will also be recorded. The trial is expected to be conducted in Shuange-Ho hospital, Taipei Medical University.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease, age between 45-80 years old.
2. With mild cognitive impairment or dementia (Clinical Dementia Rating Scale >= 0.5)

Exclusion Criteria:

- People who have

1. pre-existing and active major neurological diseases other than PD
2. with a previous history of seizures
3. with implanted metallic objects that would contraindicate rTMS
4. unable to perform fMRI
5. with skin damage on the stimulation area
6. with multiple sclerosis
7. with large ischemic scars
8. with a family history or medical history of seizures, epilepsy
9. brain damage may affect the threshold for inducing epilepsy
10. taken tricyclic antidepressants, analgesics, or anything that may lower the threshold for inducing epilepsy
11. with sleep disorders during the rTMS treatment
12. with severe alcohol abuse or use of epilepsy drugs
13. with severe heart disease or uncontrollable migraine caused by high intracranial pressure
14. who are actively suicidal during the trial period, have recurring major medical disorders, or with neurological co-morbidities such as space occupying lesions, CVA, aneurysms etc

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Mini-Mental State Examination (MMSE) score at 1 months after theta burst stimulation | Baseline and 1 months after theta burst stimulation
  Measure score change on Mini-Mental State Examination. The maximum score is 30 and the minimum score is 0, with higher score means better outcome.
Change from baseline Wechsler Memory Scale (WMS) score at 1 months after theta burst stimulation | Baseline and 1 months after theta burst stimulation
  Measure score change on Wechsler Memory Scale (WMS). Higher score means better outcome.
Change from baseline Trial Making Test A and B at 1 months after theta burst stimulation | Baseline and 1 months after theta burst stimulation
  Measure score change on Trial Making Test A and B
Change from baseline Category Fluency Test at 1 months after theta burst stimulation | Baseline and 1 months after theta burst stimulation
  Measure score change on Category Fluency Test
Change from baseline Clock Drawing Test at 1 months after theta burst stimulation | Baseline and 1 months after theta burst stimulation
  Measure score change on Clock Drawing Test

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Tai Chien-Tai, MD, PHD, Study Chair — Shuang Ho hospital, Taipei Medical University
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Some of the participants hesitate to share IPD.